CLINICAL TRIAL: NCT01626482
Title: Effect of Kinesio Tape in Muscle Fatigue Measured by Biering-Sorensen Test
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEU-003
Record Dates: First submitted 2012-06-15; First posted 2012-06-22 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Bandages

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Sham tape (Placebo Comparator)
  Interventions: Other: Placebo
- Kinesio Tape (Experimental)
  Interventions: Other: Kinesio Taping

INTERVENTIONS:
Other: Kinesio Taping — The taping consisted of two strips of material in the form of "I" on both sides of the lumbar spine, from the sacroiliac joint to the ipsilateral transverse process of D12.
  Other Names: Bandage
  Arms: Kinesio Tape
Other: Placebo — The placebo taping consisted of two 10 cm length strips of the same material, adhered transversely to the skin of the paravertebral muscles fibers
  Arms: Sham tape

SUMMARY:
Muscle fatigue affects adversely the athletes´ performance and it is therefore one of the most investigated topics currently. However we do not know accurately the mechanisms that produce it.

The aim of this study is to determine the influence of the Kinesio taping (KT) application in the paravertebral muscle fatigue in a sample of healthy young subjects.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years
* They were motivated to be included in the study

Exclusion Criteria:

* History of Low Back Pain (LBP) in the last 6 months that had lasted for at least 1 week and / or had required medical attention and / or had been off sick
* Back surgery
* Been diagnosed with cardiovascular disease or neurological or herniations, protrusions or severe scoliosis
* Had pain from a disease presenting infection, tumor or injury of an anatomical structure involved in the test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Time of maintenance in the Biering-Sorensen Test | Seconds
  Duration in seconds of the Biering-Sorensen Test

CONTACTS AND LOCATIONS:
Locations (1):
- San Pablo CEU University, Boadilla del Monte, Madrid, Spain